CLINICAL TRIAL: NCT04369313
Title: Effect of Delayed Cord Clamping on Neonatal Jaundice and Blood Gas Analysis in Infants Born to Gestational Diabetes Mellitus Mothers
Brief Title: Effect of DCC on Neonatal Jaundice and Blood Gas Analysis in Infants Born to GDM Mothers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SAHoWMU-CR2020-07-107
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Gestational Diabetes Mellitus; Neonatal Hyperbilirubinemia; Neonatal Asphyxia
MeSH Terms: conditions — Diabetes, Gestational; Hyperbilirubinemia, Neonatal; Asphyxia Neonatorum | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- delayed cord clamping (Experimental): clamping the cord at least 30s at birth
  Interventions: Procedure: delayed cord clamping
- early cord clamping (Other): umbilical cord clamping before 15 seconds
  Interventions: Procedure: early cord clamping

INTERVENTIONS:
Procedure: delayed cord clamping — umbilical cord clamping more than 30 seconds after birth
  Arms: delayed cord clamping
Procedure: early cord clamping — umbilical cord clamping within 15 seconds after birth
  Arms: early cord clamping

SUMMARY:
Evidence for benefited newborns following delayed cord clamping (DCC), including increasing hemoglobin and hematocrit levels, improving iron stores, and decreasing need for blood transfusion and incidence of intraventricular hemorrhage, in term or preterm infants led the American College of Obstetricians and Gynecologists (ACOG) to recommend a delayed cord clamping at least 30-60 seconds in vigorous term and preterm infants at birth. Although DCC has been found to be beneficial to infants, the additional blood provided by DCC could increase the incidence of jaundice that requires phototherapy and the hyperbilirubinemia, and the time prolonged by DCC might jeopardize timely resuscitation efforts, if needed. The acid-base status in umbilical cord blood at birth reflects the newborn's aerobic and anaerobic intrauterine metabolisms and is an objective measure of the fetal exposure and response to hypoxia during labour.

Gestational diabetes mellitus (GDM) is a condition in which glucose intolerance develops during pregnancy. It has been estimated in 2009 that nearly 7% of pregnancies are complicated by diabetes and approximately 86% of these cases represented women with GDM. The Hyperglycemia and Adverse Pregnancy Outcome study (HAPO) revealed that the infants of diabetic mothers (IDMs) are at increased risk of neonatal hypoglycemia, hyperbilirubinemia, shoulder dystocia, and birth trauma. And newborns to diabetic mothers are at increased risk of neonatal respiratory distress syndrome (RDS) and hypoxia, a major cause of admission in neonatal intensive care units. There is little direct evidence on the implementation of delayed umbilical cord clamping in the risk group of IDMs. Therefore, it no clear that the effectiveness and impairment of DCC in IDMs.

Therefore, the investigators conducted a prospective study in performing DCC in the infants of diabetic mothers versus the newborns with early cord clamping (ECC) to assess the effect of DCC on neonatal bilirubin levels, hyperbilirubinemia incidence, acid-base status and hypoxia in IDMs.

ELIGIBILITY:
Inclusion Criteria:

People in the study should meet the following inclusion criteria:

* Must be a singleton pregnancy
* Clinical diagnosis of gestational diabetes mellitus according to ACOG Practice Bulletin

Exclusion Criteria:

* Pregnant women and neonates were excluded if they met the exclusion criteria (not included in if meeting one of following items )
* Maternal clinical diseases (hypertension disorders, abnormal liver function, Rhesus negative blood group or other blood system disease)
* Maternal other pregnancy complications (polyhydramnios, oligohydramnios, placenta praevia, and abruptio placentae).
* Delivery before 37 weeks or after 42 weeks
* Neonatal weight was < 2.5 kg or>4.0 kg
* Neonates had major congenital malformations (congenital anal atresia, congenital biliary atresia, congenital heart disease and so on, whether prenatal suspicion or diagnosis postpartum)
* Neonatal septicemia, hemolytic disease or other diseases affecting bilirubin metabolism.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 70 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
neonatal cord acid-base status | within the 15 minutes after delivery
  arterial cord samples were analyzed within 15 min by blood gas analyzer
neonatal transcutaneous bilirubin level | within the 1 to 3 days of age
  The transcutaneous bilirubin was measured by the uniform TcB device three times a day
Number of infants with neonatal jaundice requiring phototherapy | within the 1 to 3 days of age
  the infants need phototherapy because of high bilirubin level
Number of infants with neonatal hyperbilirubinemia | within the 1 to 3 days of age
  the infants need phototherapy because of high bilirubin level

SECONDARY OUTCOMES:
neonatal initial blood glucose levels | within the 30 minutes after delivery
  The initial blood glucose levels were measured within 30 minutes after birth and before breastfeeding

CONTACTS AND LOCATIONS:
Locations (1):
- department of obstetrics of Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Zhao X, Xu A, Lu X, Chen B, Hua Y, Ma Y. Association of phthalates exposure and sex steroid hormones with late-onset preeclampsia: a case-control study. BMC Pregnancy Childbirth. 2024 Sep 3;24(1):577. doi: 10.1186/s12884-024-06793-5. PMID 39227873
- [Derived] Pan S, Lu Q, Lan Y, Peng L, Yu X, Hua Y. Differential effects of delayed cord clamping on bilirubin levels in normal and diabetic pregnancies. Eur J Pediatr. 2022 Aug;181(8):3111-3117. doi: 10.1007/s00431-022-04536-2. Epub 2022 Jun 25. PMID 35751710
- [Derived] Shao H, Lan Y, Qian Y, Chen R, Peng L, Hua Y, Wang X. Effect of later cord clamping on umbilical cord blood gas in term neonates of diabetic mothers: a randomized clinical trial. BMC Pediatr. 2022 Mar 1;22(1):111. doi: 10.1186/s12887-022-03170-z. PMID 35232426